CLINICAL TRIAL: NCT03645200
Title: Fluzoparib Combined With Apatinib for the Treatment of Carrying TP53 Harmful Mutations in Advanced Refractory Solid Tumors of the I Stage Clinical Study
Brief Title: Treatment of Carrying TP53 Harmful Mutations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP53MuToma
Record Dates: First submitted 2018-08-22; First posted 2018-08-24 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2018-08

CONDITIONS: Advanced Cancer
Keywords: TP53; Solid tumor; Fluzoparib; Apatinib
MeSH Terms: interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib combined with Apatinib (Experimental): Fluzoparib in the initial dose of 40mg.bid started into the group of participants, group A combined with a fixed dose of Apatinib 250mg.qd for treatment, followed by the 40mg.bid, 60mg.bid, 80mg.bid, 100mg.bid dose increase.
  Fluzoparib in the initial dose of 40mg.bid started into the group of participants, Group B was treated with a fixed dose of Apatinib 500mg.qd, followed by an increase in doses of 40mg.bid, 60mg.bid, 80mg.bid, 100mg.bid .
  Interventions: Drug: Fluzoparib combined with Apatinib

INTERVENTIONS:
Drug: Fluzoparib combined with Apatinib — Fluzoparib :
  40mg.bid, morning and evening each time, interval of 12 hours or so, the first oral administration 72 hours later
  Apatinib :
  250mg or 500mg take one day, 72 hours later, the continuous drug delivery phase (B-C1D1) was entered into the Fluzoparib, that is, the Fluzoparib capsule with 40mg.bid, every morning and evening, each time, interval of 12 hours, the Apatinib tablets daily with the Fluzoparib capsule with the same service, fixed doses of 250mg or 500mg, daily. Continuous drug delivery for 28 days for one cycle
  Other Names: Apatinib mesylate tablets

SUMMARY:
Assessment of the safety and tolerability of Fluzoparib combined with Apatinib in the treatment of advanced refractory solid tumors with TP53 harmful mutations.

DETAILED DESCRIPTION:
Results of the clinical trial of the combination of Fluzoparib and Apatinib in the treatment of gastric cancer animal model and the drug PARP inhibitor alone, PARP inhibitor combined with VEGFR inhibitor, Patients with advanced refractory solid tumors with TP53 harmful mutations can be expected to be safe and effective in the treatment of Fluzoparib and Apatinib.

ELIGIBILITY:
Inclusion Criteria:

* Age is 18≥years ≤70 years .
* ECOG body State is 0~1 score.
* The estimated survival period are greater than 3 months .
* Histologic or cytological diagnosis of advanced refractory tumors that are ineffective or without standard treatment by standard multi-line therapy. The definition of treatment invalidity: progression of disease after multiple line therapy.
* With the relevant qualification agencies NGS (second generation sequencing) report, and the molecular Oncology Expert Committee identified TP53 as the main harmful mutation.
* The patient has at least one measurable lesion that can be assessed by CT or MRI (RECIST 1.1).
* Previous treatment of any anti-tumor therapy (including radiotherapy, chemotherapy, hormone therapy, surgery, or molecular targeting therapy) ended with the Thou Yan ≥4 weeks (to the first medication) in this trial.
* Urine routine display urine protein <2+, if urine protein qualitative ≥2+, should accept 24 hour urine protein quantitative detection, ≤ 1g can be entered into a group.
* Good organ function level ( no blood transfusion, no use of G-CSF in the first 7 days of screening ; no drug correction;7 days without loss ALB):ANC≥ 1.5x109/L;WBC≥ 3x109 /L;PLT≥80x109/L ;Hb≥90g/l; TBIL≤1.5xULN;ALT and AST≤2.5xULN; ALB≥29g/l ;BUN and Cr ≤1. 5xULN ;LVEF ≥50%;Fridericia method to correct QT Inter-period (QTcF ) Male <450 ms , Women <470 ms .
* Women of childbearing age are required to take effective contraceptive measures at least 8 weeks after taking part in the study and after the last drug delivery .
* Can follow the test plan according to the judgment of the investigator.
* Volunteer to participate in this clinical trial, have the ability to understand the research requirements, can give written informed consent.

Exclusion Criteria:

* Anticancer drugs, including Fluzoparib that used or were using PARP as a target.
* Antineoplastic agents used or using VEGFR targets, including Apatinib.
* As a participant in the clinical trial, and the signing of the informed consent of the last clinical trial at the end of the interval of less than days.
* Has a blood system-related tumor.
* Receive any anti-tumor treatment (including radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeting therapy) within 4 weeks before delivery;
* Double phosphate drug treatment was received in the first 4 weeks of the drug delivery;
* There is a CTCAE grade II toxicity caused by previous treatment.
* Hypertension is not controlled (systolic pressure is greater than 150mmHg, or diastolic pressure is greater than 90 mmHg); or a history of congestive heart failure (American Heart Association heart function grade ≥2 Level).
* Clinically significant heart disease, including but not limited to: congestive heart failure, symptomatic coronary artery disease, arrhythmia, myocardial infarction, QTc period ≥470ms.
* Intestinal obstruction or CTCAE 3 or 4 upper digestive tract bleeding in the first 4 weeks before the drug delivery.
* Inability to swallow, inflammatory bowel disease or uncontrollable nausea, vomiting, diarrhea or other gastrointestinal disorders that seriously affect drug use and absorption.
* The tumor metastasis of central nervous system was diagnosed by the researchers.
* A history of severe venous thrombosis or pulmonary embolism.
* There is a third interstitial fluid (such as large pleural effusion and ascites) that cannot be controlled by drainage or other means.
* There is still an electrolyte disorder that cannot be corrected when the group is given a drug.
* In the first 7 days before the group received a strong CYP3A4 inhibitor treatment, or in the first day of the group received a strong effect CYP3A4 Inducer therapy.
* Active HBV, HCV infection (HBV copy number ≥104 copies/ml, the number of copies of HCV virus ≥103 copies /ml).
* There is a history of immune deficiency, including HIV testing positive, or other acquired, congenital immunodeficiency disease, or a history of organ transplantation.
* Pregnancy, breast-feeding female patients.
* In patients with bone metastases, palliative radiotherapy (radiotherapy area,5% bone marrow region) was received within 4 weeks before the group's entry.
* According to the researchers ' judgment, there are serious, uncontrollable risks to patients ' safety, or associated diseases (such as severe diabetes, thyroid disease, infection, spinal cord compression, superior vena cava syndrome, neurological or psychiatric disorders) that affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Dosage (provide right dosage for II phase clinical trial) | 12 months
  provide right dosage for II phase clinical trial

SECONDARY OUTCOMES:
ORR: objective response rate | 12 months
  objective response rate
DCR: disease control rate | 12 months
  disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Haitao Wang, Ph.D, Principal Investigator — Tianjin Medical University Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China